CLINICAL TRIAL: NCT07066280
Title: Skin Repairing Cream for the Prevention of Radiation Dermatitis and Regulation of Skin Microbial Environment in Breast Cancer: A Multicenter, Prospective, Randomized Controlled Study
Brief Title: Modulating the Skin Microbiome to Prevent Radiation Dermatitis in Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SYSKY-2024-1129-01
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-03

CONDITIONS: Skin Microbiome; Breast Cancer; Radiation Dermatitis
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: Skin Repairing Cream
- Control group (Other)
  Interventions: Other: Cetaphil® Moisturizing Cream as Inactive Control

INTERVENTIONS:
Drug: Skin Repairing Cream — Skin Repairing Cream containing natural weak-acid
  Arms: Experimental group
Other: Cetaphil® Moisturizing Cream as Inactive Control — Cetaphil® Moisturizing Cream
  Arms: Control group

SUMMARY:
Acute radiation dermatitis (ARD) is the most common treatment-related adverse reaction following radiotherapy after modified radical mastectomy and/or prosthetic breast reconstruction in breast cancer patients. Moderate-to-severe ARD may compromise cosmetic outcomes and quality of life, and even impair radiotherapy efficacy. Current pharmacological prophylactic measures clinically employed - including topical corticosteroids, superoxide dismutase, and trolamine cream - demonstrate suboptimal efficacy and lack high-level evidence-based medical support. Emerging research indicates an association between cutaneous microbial homeostasis and ARD development, suggesting that maintaining skin surface acidity and modulating microecological balance may represent more effective preventive strategies.

This study evaluates the efficacy and safety of a natural weak-acid macromolecular/small molecular repair cream in preventing ARD among post-operative breast cancer patients receiving radiotherapy through skin microbiome modulation. We enrolled 326 high-risk early-stage breast cancer patients scheduled for post-operative radiotherapy and randomized them to compare the superiority of the natural weak-acid repair cream versus conventional care with moisturizer. Concurrent skin microbiome sampling was performed to assess microecological changes and their impact on ARD development. The findings will provide high-level clinical evidence and theoretical basis for the safer and more effective application of this natural weak-acid repair cream in preventing post-radiotherapy ARD in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and <70 years, with pathologically confirmed breast cancer;

  * TNM stage T1-3N1-3M0 or T3-4N0M0;

    * Underwent mastectomy with or without implant reconstruction; ④ Medically fit for adjuvant radiotherapy (i.e., in good general condition to tolerate expected side effects such as fatigue, nausea, or vomiting); ⑤ No concurrent use of other skincare products throughout the study period;

      * Voluntary participation with signed informed consent, agreeing to comply with investigator-directed use of the trial product.

Exclusion Criteria:

* Prior history of radiotherapy;

  * Severe systemic diseases (e.g., significant cardiac, hepatic, or renal dysfunction; immunocompromising conditions such as lymphoma, acquired immunodeficiency syndrome [AIDS], or Wiskott-Aldrich syndrome) or history of other malignancies; ③ Skin reactions due to systemic therapies (e.g., chemotherapy, immunotherapy) or active dermatologic conditions in the treatment area;

    * Known hypersensitivity to the natural weak-acid macromolecular/small molecular repair cream or any of its components; ⑤ Current participation in other clinical trials or participation within the past 3 months, or judged by investigators to have poor compliance that would prevent completion of the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 326 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute radiation dermatitis (ARD) of grade 2-5 | Before RT and within two weeks of completion of RT

SECONDARY OUTCOMES:
quality of life (QoL) | Before RT and within two weeks of completion of RT
  Quality of Life assessment using the Skindex-16 questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No